CLINICAL TRIAL: NCT02579941
Title: Evaluation of the Minimum Concentration of Tranexamic Acid Required to Inhibit Fibrinolysis in a Population of Pregnant Women at Term.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Philippe VAN DER LINDEN, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUB-Fibrinolyse
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Hyperfibrinolysis
Keywords: Hyperfibrinolysis; Pregnant women at term; Tranexamic acid
MeSH Terms: interventions — Blood Specimen Collection; Gravidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pregnant women at term, vaginal childbirth (Experimental)
  Interventions: Procedure: Blood sampling (pregnant)
- Pregnant women at term, cesarean delivery (Experimental)
  Interventions: Procedure: Blood sampling (pregnant)
- Female volunteers, age 18 to 40 (Experimental)
  Interventions: Procedure: Blood sampling (non pregnant)

INTERVENTIONS:
Procedure: Blood sampling (pregnant) — 5.4 ml of venous blood will be taken during the delivery or the caesarian procedure, in addition to the standard of care blood sampling.
  This blood vial will be sent to the coagulation laboratory and all tests will be performed in vitro. The blood sample will be split in several aliquots. In each blood sample, fibrinolysis will be activated by the plasminogen tissular activator (tPA - concentration: 1066 UtPA/ml). Tranexamic acid will be added at increasing concentrations (2.5 microg/ml up to 40 microg/ml) to each sample and coagulation will be measured by two different tests: EXTEM and NATEM.
  Arms: Pregnant women at term, cesarean delivery; Pregnant women at term, vaginal childbirth
Procedure: Blood sampling (non pregnant) — 5.4 ml of venous blood will be taken.
  This blood vial will be sent to the coagulation laboratory and all tests will be performed in vitro. The blood sample will be split in several aliquots. In each blood sample, fibrinolysis will be activated by the plasminogen tissular activator (tPA - concentration: 1066 UtPA/ml). Tranexamic acid will be added at increasing concentrations (2.5 microg/ml up to 40 microg/ml) to each sample and coagulation will be measured by two different tests: EXTEM and NATEM.
  Arms: Female volunteers, age 18 to 40

SUMMARY:
Pregnancy induces a physiological change of hemostasis to a prothrombotic state : protein S decrease and increase of virtually all the clotting factors, in particular fibrinogen, von Willebrand factor and factor VIII. However, a state of hyperfibrinolysis may occur in the immediate postpartum period (especially after placental delivery), thereby promoting postpartum hemorrhage.

This state of hyperfibrinolysis is associated with the use of transfusions of blood products and the realization of hysterectomy.It is currently the most common etiology of maternal mortality in childbirth.There is an imperative to develop an efficient and reliable protocol for the management of this postpartum complication.

Tranexamic acid is an anti-fibrinolytic agent (like lysine) which acts by preventing the conversion of plasminogen to plasmin, by blocking the binding of plasminogen to the heavy chain of fibrin.The optimal dose of tranexamic acid enabling to inhibit fibrinolysis without increasing the complications rate remains to be defined. It is in this context that the investigators aim to evaluate, in an in-vitro model, the minimum dose of tranexamic acid required to inhibit fibrinolysis after activation of the latter by t-PA. The degree of fibrinolysis will be evaluated by thromboelastometry.

DETAILED DESCRIPTION:
Pregnancy induces a physiological change of hemostasis to a prothrombotic state : protein S decrease and increase of virtually all the clotting factors, in particular fibrinogen, von Willebrand factor and factor VIII. However, a state of hyperfibrinolysis may occur in the immediate postpartum period (especially after placental delivery), thereby promoting postpartum hemorrhage.

This state of hyperfibrinolysis is associated with the use of transfusions of blood products and the realization of hysterectomy.It is currently the most common etiology of maternal mortality in childbirth. Although its incidence is low in western countries, it remains very high in the world.There is an imperative to develop an efficient and reliable protocol for the management of this postpartum complication.

Tranexamic acid is an anti-fibrinolytic agent (like lysine) which acts by preventing the conversion of plasminogen to plasmin, by blocking the binding of plasminogen to the heavy chain of fibrin.The use of this agent has spread in recent years in many types of surgery (cardiac, orthopedic, etc.), and in patient polytrauma. However, the number of studies evaluating its efficacy in the management (treatment and / or prevention) of postpartum hemorrhage is limited. In addition, the doses used are extrapolated from studies of a different population (multiple trauma, cardiac surgery, etc).

The tranexamic acid proposed scheme is currently used is not suitable for the population of pregnant women at term. It was established arbitrarily on the basis of the adult population without considering the physiological and metabolic characteristics of the term pregnancy. The optimal dose of tranexamic acid enabling inhibition of fibrinolysis, without increasing the complications rate, remains thus to be defined.

It is in this context that the investigators aim to evaluate, in an in-vitro model, the minimum dose of tranexamic acid required to inhibit fibrinolysis after activation of the latter by t-PA. The degree of fibrinolysis will be evaluated by thromboelastometry.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women group:

* pregnant women at term (>37 weeks of gestation)
* patients admitted for delivery or elective cesarian section
* written informed consent

Healthy volunteers group:

- women aged from 18 to 40

Exclusion Criteria:

* Dying patients (ASA 5)
* Jehovah's witnesses
* Patients with pre-eclampsia, HELLP syndrome, placenta previa or placental abruption.
* Multiple pregnancy
* Presence of preoperative coagulation disorders defined as: platelets <150,000 / mm3; PTT <70%; aPTT> 33 sec; fibrinogen <350 mg / dL.
* Treatment with anticoagulant or antiplatelet agent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Coagulation (EXTEM) | within 24h of blood collection
  Coagulation will be tested using the EXTEM test (test evaluating the extrinsic coagulation pathway after its activation by tissue factor)
Coagulation (NATEM) | within 24h of blood collection
  Coagulation will be tested using the NATEM test (test evaluating coagulation after startem addition (for recalcification of citrated blood) and without activator addition)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van der Linden, MD, Principal Investigator — CHU Brugmann; Arnaud Lechien, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Cerneca F, Ricci G, Simeone R, Malisano M, Alberico S, Guaschino S. Coagulation and fibrinolysis changes in normal pregnancy. Increased levels of procoagulants and reduced levels of inhibitors during pregnancy induce a hypercoagulable state, combined with a reactive fibrinolysis. Eur J Obstet Gynecol Reprod Biol. 1997 May;73(1):31-6. doi: 10.1016/s0301-2115(97)02734-6. PMID 9175686
- [Background] Bonnar J, McNicol GP, Douglas AS. Coagulation and fibrinolytic mechanisms during and after normal childbirth. Br Med J. 1970 Apr 25;2(5703):200-3. doi: 10.1136/bmj.2.5703.200. PMID 5443405
- [Background] Brenner B. Haemostatic changes in pregnancy. Thromb Res. 2004;114(5-6):409-14. doi: 10.1016/j.thromres.2004.08.004. PMID 15507271
- [Background] Faraoni D, Carlier C, Samama CM, Levy JH, Ducloy-Bouthors AS. [Efficacy and safety of tranexamic acid administration for the prevention and/or the treatment of post-partum haemorrhage: a systematic review with meta-analysis]. Ann Fr Anesth Reanim. 2014 Nov;33(11):563-71. doi: 10.1016/j.annfar.2014.07.748. Epub 2014 Oct 18. French. PMID 25450729
- [Background] Sentilhes L, Lasocki S, Ducloy-Bouthors AS, Deruelle P, Dreyfus M, Perrotin F, Goffinet F, Deneux-Tharaux C. Tranexamic acid for the prevention and treatment of postpartum haemorrhage. Br J Anaesth. 2015 Apr;114(4):576-87. doi: 10.1093/bja/aeu448. Epub 2015 Jan 8. PMID 25571934
- [Background] Ronsmans C, Graham WJ; Lancet Maternal Survival Series steering group. Maternal mortality: who, when, where, and why. Lancet. 2006 Sep 30;368(9542):1189-200. doi: 10.1016/S0140-6736(06)69380-X. PMID 17011946
- [Background] Ortmann E, Besser MW, Klein AA. Antifibrinolytic agents in current anaesthetic practice. Br J Anaesth. 2013 Oct;111(4):549-63. doi: 10.1093/bja/aet154. Epub 2013 May 9. PMID 23661406
- [Background] Collis RE, Collins PW. Haemostatic management of obstetric haemorrhage. Anaesthesia. 2015 Jan;70 Suppl 1:78-86, e27-8. doi: 10.1111/anae.12913. PMID 25440400